CLINICAL TRIAL: NCT01948219
Title: An Evaluation of the ENTegral Artificial Larynx (AL) in Patients Indicated for Total Laryngectomy
Brief Title: ENTegral Artificial Larynx Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: ProTiP Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LA-01-PEC-1
Record Dates: First submitted 2013-09-16; First posted 2013-09-23 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Total Laryngectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ENTegral Artificial Larynx implant (Experimental): ENTegral Artificial Larynx implantation
  Interventions: Device: ENTegral Artificial Larynx implant

INTERVENTIONS:
Device: ENTegral Artificial Larynx implant

SUMMARY:
The objective of this clinical study is to evaluate the feasibility, safety and efficacy of the ENTegral Artificial Larynx (AL) in patients indicated for total laryngectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age more than or equal to 18 years old
* Is indicated for total laryngectomy (first intention)
* Must be able to comply with study requirements
* Must be able to understand and be willing to provide written informed consent

Exclusion Criteria:

* Any condition that precludes the implantation of the ENTegral AL
* Existing coagulation disorder
* Contraindication for general anesthesia
* Tumoral extension outside of the larynx invading through extra-laryngeal structures
* Previous radiotherapy
* Life-expectancy < 12 months
* Be pregnant of breastfeeding or intention to becoming pregnant during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of device implant procedure | 1 year
  Number of patients with adverse event associated with device implantation procedure

OTHER OUTCOMES:
Quality of life | 1, 3, 6 months and 1 year
  Quality of life using EORTC QLQ-C30 and QLQ-H&N25 questionnaires
Number of patients with adverse events | 1 year
  Number of patients with adverse events will be assessed at each follow-up during the 1 year patient follow-up
Dyspnea evolution | 1,2,3,6,9 months and 1 year
  Dyspnea evaluation using the Heyse-Moore scale at 1, 2, 3, 6, 9 months and 1 year
Phonation evolution | 1,2,3,6,9 months and 1 year
  Patient phonation (able to talk and be understood, whispered voice) will be assessed at 1, 2, 3, 6, 9 months and 1 year
Implant use | 1,2,3,6,9 months and 1 year
  Implant use (manual closure of the tracheostomy orifice) duration will be assessed at 1, 2, 3, 6, 9 months and 1 year, allowing eventually to surgically close the orifice

CONTACTS AND LOCATIONS:
Locations (3):
- CHU Mont-Godinne, Yvoir, Belgium
- France (2):
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse